CLINICAL TRIAL: NCT00662545
Title: Entecavir Intensification for Persistent Hepatitis B Virus (HBV) Viremia in HIV-HBV Infection
Brief Title: Entecavir Intensification for Persistent HBV Viremia in HIV-HBV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A109324; AI463-162
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections; Hepatitis B
Keywords: HIV; Hepatitis B; treatment experienced
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — entecavir; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Racivir; Lamivudine; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Entecavir 1 mg for 24 weeks in addition to continued standard of care antiretroviral therapy containing tenofovir in addition to emtricitabine or lamivudine
  Interventions: Drug: Entecavir with continued standard of care antiretroviral therapy
- B (Active Comparator): continued standard of care antiretroviral therapy which will include tenofovir in addition to emtricitabine or lamivudine
  Interventions: Drug: continued standard of care with tenofovir in addition to emtricitabine or lamivudine

INTERVENTIONS:
Drug: Entecavir with continued standard of care antiretroviral therapy — 1 mg by mouth daily
  Other Names: Baraclude, Tenofovir, Truvada, Viread, 3TC, FTC, Epivir, Emtriva
  Arms: A
Drug: continued standard of care with tenofovir in addition to emtricitabine or lamivudine — continued standard of care with tenofovir in addition to emtricitabine or lamivudine
  Other Names: Tenofovir, Truvada, Viread, 3TC, FTC, Epivir, Emtriva
  Arms: B

SUMMARY:
This study will evaluate HIV-HBV infected individuals who have evidence of HBV replication in the blood after taking 48 weeks of more of the HBV active medication tenofovir in combination with emtricitabine or lamivudine. Eligible participants will be randomized to receive 24 weeks of entecavir (ETV) 1 mg versus continued standard of care antiretroviral therapy. After 24 weeks, individuals on entecavir or who remain HBV viremic on standard of care will receive ETV o for an additional 24 weeks. The hypothesis is that intensification with entecavir will reduce HBV DNA at 24 weeks more than continued antiretroviral therapy without entecavir.

DETAILED DESCRIPTION:
Design: This is a randomized, controlled pilot study of open-label entecavir for the treatment of persistent HBV viremia in HIV-HBV coinfected individuals who have failed to suppress HBV replication after 48 weeks on tenofovir containing therapy.

Primary Objective: To evaluate the mean log reduction of HBV DNA with entecavir(ETV) intensification in comparison to continued standard therapy with tenofovir and lamivudine/emtricitabine at 24 weeks of therapy

Study Population: HIV-HBV co-infected individuals with detectable HBV DNA after 48 weeks of therapy with tenofovir and lamivudine/emtricitabine whose HIV viremia is well controlled ( < 75 copies at time of enrollment)

Treatment: Subjects will be randomized to continue with standard therapy or to receive intensification with 1 mg daily of open label entecavir for the 24 week duration of the study.

Sample Size: 24 subjects will be enrolled.

Duration 24 weeks of treatment

Primary Endpoint: Mean log10 reduction of HBV DNA at 24 weeks of standard therapy vs. entecavir intensification.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* HIV infection, documented in patient medical record. Acceptable forms of documentation include positive HIV antibody or detectable HIV RNA.
* Chronic HBV infection, defined as HBsAg positivity. Both hepatitis B "e" antigen (HBeAg) positive and negative subjects will be eligible.
* Detectable HBV DNA ( > 160 copies/ml) after 48 weeks of therapy with TDF in conjunction with either 3TC or FTC
* Compensated liver disease, defined as a Child-Pugh-Turcot(CPT) Score <7 at the time of enrollment.

Note: If Bilirubin in elevated, direct and indirect bilirubin levels will be evaluated. If only indirect bilirubin elevated, direct bilirubin will be used for CPT score. If BOTH direct and indirect bilirubin are elevated, total bilirubin will be used for the CPT score.

* Stable antiretroviral therapy with no changes in the prior 8 weeks due to antiretroviral failure. HIV therapy modification for reasons other than virologic failure and without change in the tenofovir(TDF), lamivudine(3TC) or emtricitabine(FTC) moiety of the antiretroviral therapy will be permitted. HIV therapy must include TDF in conjunction with 3TC or FTC, and at least one other anti-HIV agent.
* HIV RNA of <75 copies/ml within 8 weeks of study enrollment.
* Estimated creatinine clearance by Cockcroft-Gault of ≥ 50 ml/min
* Serum alpha-fetoprotein (AFP) of ≤50 ng/ml within 8 weeks of study entry, or if elevated > 50 ng/ml, an imaging study demonstrating no evidence of hepatic tumor within 8 weeks of enrollment.
* Female study volunteers must not participate in a conception process (e.g., active attempt to become pregnant). If participating in sexual activity that could lead to pregnancy, the female study volunteer must use the following forms of contraception while receiving study-specific medication(s) and for 30 days after stopping the medication. One of the following methods MUST be used appropriately:

  * Condoms1 (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * intrauterine device(IUD)
  * Hormonal-based method

    1. Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission.

Note: Subjects with concomitant Hepatitis C infection will be permitted to enroll.

Exclusion Criteria:

* Allergy or sensitivity to study drug
* Pregnancy, breastfeeding or unwillingness/inability to adhere to contraceptive methods for the duration of the study
* Prisoners or subjects who are incarcerated.
* Evidence of malignancy that would make the subject, in the opinion of the investigator, unsuitable for the study. This includes any systemic antineoplastic or immunomodulatory treatment or radiation within 24 weeks prior to study entry or the expectation that such treatment will be needed at any time during the study.
* Receipt of systemic corticosteroids within 90 days prior to study entry (as this medication may increase HBV replication).
* Investigational anti-HIV agents will be allowed on a case-by-case basis with the approval of the protocol team.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Any active medical, psychiatric or social circumstance that in the opinion of the investigator puts the subject at potential risk from study participation or makes adherence to the study protocol unlikely.
* Receipt of the following drugs with anti-HBV activity within 90 days prior to study entry or anticipated receipt during the course of the study including: adefovir(ADV), telbivudine, alpha interferon, penciclovir (Denavir) (except if given for < 4 weeks), famciclovir (Famvir), diaminopurine dioxolane (DAPD), clevudine (L-FMAU), thymosin alpha 1, ganciclovir (treatment limited to < 7 days is acceptable) (Cytovene), L-deoxythymidine, and L-deoxythymidine compounds and other investigational agents with anti-HBV activity.
* Receipt of nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, vancomycin, cidofovir [Vistide], foscarnet [Foscavir], cisplatin, intravenous pentamidine [Pentam], oral tacrolimus [Prograf], cyclosporine [Sandimmune]) or the competitor of renal excretion, probenecid (Benemid), within 8 weeks prior to study entry or expected use of these agents during the course of the study. (Topical tacrolimus is allowed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne F Luetkemeyer, MD, Principal Investigator — HIV/AIDS Division, San Francisco General Hospital, University of California, San Francisco
Locations (1):
- San Francisco General HIV Clinical Trials Group, San Francisco, California, United States

REFERENCES:
- [Background] Thio CL, Seaberg EC, Skolasky R Jr, Phair J, Visscher B, Munoz A, Thomas DL; Multicenter AIDS Cohort Study. HIV-1, hepatitis B virus, and risk of liver-related mortality in the Multicenter Cohort Study (MACS). Lancet. 2002 Dec 14;360(9349):1921-6. doi: 10.1016/s0140-6736(02)11913-1. PMID 12493258
- [Background] Konopnicki D, Mocroft A, de Wit S, Antunes F, Ledergerber B, Katlama C, Zilmer K, Vella S, Kirk O, Lundgren JD; EuroSIDA Group. Hepatitis B and HIV: prevalence, AIDS progression, response to highly active antiretroviral therapy and increased mortality in the EuroSIDA cohort. AIDS. 2005 Mar 24;19(6):593-601. doi: 10.1097/01.aids.0000163936.99401.fe. PMID 15802978
- [Background] Colin JF, Cazals-Hatem D, Loriot MA, Martinot-Peignoux M, Pham BN, Auperin A, Degott C, Benhamou JP, Erlinger S, Valla D, Marcellin P. Influence of human immunodeficiency virus infection on chronic hepatitis B in homosexual men. Hepatology. 1999 Apr;29(4):1306-10. doi: 10.1002/hep.510290447. PMID 10094979
- [Background] Fattovich G, Rugge M, Brollo L, Pontisso P, Noventa F, Guido M, Alberti A, Realdi G. Clinical, virologic and histologic outcome following seroconversion from HBeAg to anti-HBe in chronic hepatitis type B. Hepatology. 1986 Mar-Apr;6(2):167-72. doi: 10.1002/hep.1840060203. PMID 3957228
- [Background] Hoofnagle JH, Shafritz DA, Popper H. Chronic type B hepatitis and the "healthy" HBsAg carrier state. Hepatology. 1987 Jul-Aug;7(4):758-63. doi: 10.1002/hep.1840070424. No abstract available. PMID 3301618
- [Background] Yu MW, Yeh SH, Chen PJ, Liaw YF, Lin CL, Liu CJ, Shih WL, Kao JH, Chen DS, Chen CJ. Hepatitis B virus genotype and DNA level and hepatocellular carcinoma: a prospective study in men. J Natl Cancer Inst. 2005 Feb 16;97(4):265-72. doi: 10.1093/jnci/dji043. PMID 15713961
- [Background] Chen G, Lin W, Shen F, Iloeje UH, London WT, Evans AA. Past HBV viral load as predictor of mortality and morbidity from HCC and chronic liver disease in a prospective study. Am J Gastroenterol. 2006 Aug;101(8):1797-803. doi: 10.1111/j.1572-0241.2006.00647.x. Epub 2006 Jun 30. PMID 16817842
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Background] Stephan C, Berger A, Carlebach A, Lutz T, Bickel M, Klauke S, Staszewski S, Stuermer M. Impact of tenofovir-containing antiretroviral therapy on chronic hepatitis B in a cohort co-infected with human immunodeficiency virus. J Antimicrob Chemother. 2005 Dec;56(6):1087-93. doi: 10.1093/jac/dki396. Epub 2005 Nov 3. PMID 16269552
- [Background] Benhamou Y, Fleury H, Trimoulet P, Pellegrin I, Urbinelli R, Katlama C, Rozenbaum W, Le Teuff G, Trylesinski A, Piketty C; TECOVIR Study Group. Anti-hepatitis B virus efficacy of tenofovir disoproxil fumarate in HIV-infected patients. Hepatology. 2006 Mar;43(3):548-55. doi: 10.1002/hep.21055. PMID 16496322
- [Background] Schmutz G, Nelson M, Lutz T, Sheldon J, Bruno R, von Boemmel F, Hoffmann C, Rockstroh J, Stoehr A, Wolf E, Soriano V, Berger F, Berg T, Carlebach A, Schwarze-Zander C, Schurmann D, Jaeger H, Mauss S. Combination of tenofovir and lamivudine versus tenofovir after lamivudine failure for therapy of hepatitis B in HIV-coinfection. AIDS. 2006 Oct 3;20(15):1951-4. doi: 10.1097/01.aids.0000247116.89455.5d. PMID 16988516
- [Background] Sheldon J, Camino N, Rodes B, Bartholomeusz A, Kuiper M, Tacke F, Nunez M, Mauss S, Lutz T, Klausen G, Locarnini S, Soriano V. Selection of hepatitis B virus polymerase mutations in HIV-coinfected patients treated with tenofovir. Antivir Ther. 2005;10(6):727-34. PMID 16218172
- [Background] Chang TT, Gish RG, de Man R, Gadano A, Sollano J, Chao YC, Lok AS, Han KH, Goodman Z, Zhu J, Cross A, DeHertogh D, Wilber R, Colonno R, Apelian D; BEHoLD AI463022 Study Group. A comparison of entecavir and lamivudine for HBeAg-positive chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1001-10. doi: 10.1056/NEJMoa051285. PMID 16525137
- [Background] Lai CL, Shouval D, Lok AS, Chang TT, Cheinquer H, Goodman Z, DeHertogh D, Wilber R, Zink RC, Cross A, Colonno R, Fernandes L; BEHoLD AI463027 Study Group. Entecavir versus lamivudine for patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1011-20. doi: 10.1056/NEJMoa051287. PMID 16525138
- [Background] Sherman M, Yurdaydin C, Sollano J, Silva M, Liaw YF, Cianciara J, Boron-Kaczmarska A, Martin P, Goodman Z, Colonno R, Cross A, Denisky G, Kreter B, Hindes R; AI463026 BEHoLD Study Group. Entecavir for treatment of lamivudine-refractory, HBeAg-positive chronic hepatitis B. Gastroenterology. 2006 Jun;130(7):2039-49. doi: 10.1053/j.gastro.2006.04.007. PMID 16762627
- [Background] McMahon MA, Jilek BL, Brennan TP, Shen L, Zhou Y, Wind-Rotolo M, Xing S, Bhat S, Hale B, Hegarty R, Chong CR, Liu JO, Siliciano RF, Thio CL. The HBV drug entecavir - effects on HIV-1 replication and resistance. N Engl J Med. 2007 Jun 21;356(25):2614-21. doi: 10.1056/NEJMoa067710. PMID 17582071
- [Background] Benhamou Y, Tubiana R, Thibault V. Tenofovir disoproxil fumarate in patients with HIV and lamivudine-resistant hepatitis B virus. N Engl J Med. 2003 Jan 9;348(2):177-8. doi: 10.1056/NEJM200301093480218. No abstract available. PMID 12519935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants recruited from medical clinic, between 7/2008 and 6/2009and 20011
Pre-assignment Details: Overall sample size was reduced to 10 due to difficulty in recruitment
Groups:
- Entecavir Intensification: Entecavir 1 mg for 24 weeks in addition to continued standard of care antiretroviral therapy containing tenofovir in addition to emtricitabine or lamivudine
- Standard of Care: continued standard of care antiretroviral therapy which will include tenofovir in addition to emtricitabine or lamivudine
Period: Overall Study
Arm/Group | Entecavir Intensification | Standard of Care
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir Intensification | Standard of Care | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
HBV DNA at enrollment [Median (Full Range); unit: log10 IU/ML] — hepatitis B DNA level
  log10 IU/ML | 3.2 [2.4 to 6.4] | 3.8 [1.9 to 7.7] | 3.2 [1.9 to 7.7]

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis B Virus (HBV) DNA
Description: HBV DNA carries the genetic blueprint of the virus. How many HBV DNA "particles" or "copies" are found in the blood indicates how rapidly the virus is reproducing in the liver.
Time Frame: week 24
Measure: Median (Full Range); unit: log 10 IU/ml
Arm/Group | Entecavir Intensification | Standard of Care
Number analyzed (Participants) | 5 | 5
log 10 IU/ml | 2.4 [0.8 to 2.41] | 0.8 [0.8 to 5.8]

2. Secondary Outcome: Incidence of Permanent Discontinuation Due to Toxicity
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Entecavir Intensification | Standard of Care
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

3. Secondary Outcome: Incidence of New Hepatic Decompensation( Ascites, Variceal Hemorrhage, Encephalopathy)
Time Frame: every 4 weeks for 24 weeks
Measure: Number; unit: participants
Arm/Group | Entecavir Intensification | Standard of Care
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

4. Secondary Outcome: Incidence of ALT Flares
Description: ALT flare: sudden increase in blood level of alanine transaminase (ALT)
Time Frame: every 4 weeks for 24 weeks
Measure: Number; unit: participants
Arm/Group | Entecavir Intensification | Standard of Care
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

5. Secondary Outcome: HIV RNA < 75 Copies/ml
Time Frame: entry, week 12, and week 24
Measure: Number; unit: participants
Arm/Group | Entecavir Intensification | Standard of Care
Number analyzed (Participants) | 5 | 5
participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Entecavir Intensification | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No